CLINICAL TRIAL: NCT02344134
Title: A Multi-center, Randomized, Double-blind Phase III Clinical Trial to Assess the Immunogenicity and Safety of NBP607 (Trivalent Inactivated Cell Culture-derived Influenza Vaccine) in Healthy Adults and Elderly Subjects
Brief Title: Study of Egg-derived Influenza Vaccine and Cell Culture-derived Influenza Vaccine in Adult and Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP607_FluA_III_2013
Record Dates: First submitted 2014-12-24; First posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2014-12

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NBP607 (Experimental): cell culture-derived trivalent inactivated subunit influenza vaccine
  Interventions: Biological: NBP607
- Agrippal S1 (Active Comparator): egg-derived trivalent inactivated subunit influenza vaccine
  Interventions: Biological: Agrippal S1

INTERVENTIONS:
Biological: NBP607 — 0.5 mL, intramuscular, a single dose
  Arms: NBP607
Biological: Agrippal S1 — 0.5 mL, intramuscular, a single dose
  Arms: Agrippal S1

SUMMARY:
The purpose of this study is to describe the immunogenicity and safety of the cell culture-derived influenza vaccine compared with the egg-derived influenza vaccine among subjects.

To describe the immunogenicity, antibody levels are evaluated by hemagglutination inhibition(HI) assay from sera obtained pre-vaccination and 21 days post-vaccination.

To describe the safety, the time of onset and duration of local and systemic solicited adverse events are assessed and reported. Unsolicited adverse events and serious adverse events are collected and categorized throughout the study period.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind study in healthy adult and elderly subjects. Subjects receive a single dose of one of the influenza vaccine formulations and provide blood samples for immunogenicity assessment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 years or older.
* The subjects who give written consent to participate in the study voluntarily and are able to comply with all study requirements.
* If female and capable of bearing children,subject has a negative urine pregnancy test result on screening and agrees to employ adequate birth control measures through the study period.

Exclusion Criteria:

* Subjects who are hypersensitive to any component of vaccine, i.e., eggs, chicken or chicken products.
* Subjects with immune deficiency disorder.
* History of Guillain-Barre syndrome.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Subjects who experienced fever within 24 hours before vaccination or with the febrile disease(exceeding 38.0℃) on screening day or with any acute respiratory infection.
* Subjects who had received immunosuppressant or immune-modifying drug within 3 months before screening.
* Subjects who had received blood products or immunoglobulin within 3 months before screening.
* Subjects who had received influenza vaccination within 6 months prior to the screening.
* Subjects who had received other vaccination within a month before screening, or those who had another vaccination scheduled within a month after study vaccination.
* Subjects who had participated in other clinical trial within 4 weeks prior to study vaccination.
* Subjects who had done blood donation within a week prior to study vaccination or planned blood donation within 7 months after study vaccination.
* Subjects with clinically significant chronic disease or malignant cancer.
* Pregnant women, breast-feeding women.
* Any other condition which, in the opinion of the Investigator, prevents the subject from participating in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1155 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMTs) for Each of the Influenza Vaccine Antigen | Day 0 and Day 21 post-vaccination
  * Percentage of Participants With Seroprotection to Each of the Influenza Vaccine Antigen Post-Vaccination.
  * Percentage of Participants Achieving Seroconversion at Day 21 Post-Vaccination With Influenza Vaccine.
  * Pre- and Post- Vaccination Geometric Mean Ratio (GMR)

SECONDARY OUTCOMES:
Immunogenicity in subjects with a pre-vaccination HI antibody titer <1:80 | Day 0 and Day 21 post-vaccination
Immunogenicity compared to control group | Day 21 post vaccination, 6 months post vaccination
Long-term Immunogenicity | 6 months post-vaccination
Percentage of participants with Solicited Local Adverse Event (AE) | During 7 days post-vaccination
Percentage of participants with Solicited Systemic Adverse Event (AE) | During 7 days post-vaccination
Percentage of participants with Unsolicited Adverse Event (AE) | During 21 days post-vaccination
Percentage of participants with Severe Adverse Event (SAE) | During 6 months post-vaccination
Vital Sign | Day 0 and Day 21 post vaccination
  Body Temperature, Blood Pressure(SBP/DBP), Pulse
Physical Examination | Day 0 and Day 21 post vaccination
  inspection, palpation (feel), percussion (tap to determine resonance characteristics), and auscultation (listen)
Clinical Laboratory Tests | Day 0 and Day 21 post vaccination
  Blood test(CBC, Coagulation, Chemistry), Urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Woojoo Kim, Principal Investigator — Korea University Guro Hospital; Seongheon Wie, Principal Investigator — Saint Vincent's Hospital, Korea; Shinwoo Kim, Principal Investigator — Kyungpook National University Hospital; Wonsuk Lee, Principal Investigator — Korea University Ansan Hospital; Jinsoo Lee, Principal Investigator — Inha University Hospital; Jacob Lee, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital; Heungjeong Woo, Principal Investigator — Dotal Sacred Heart Hospital

REFERENCES:
- [Derived] Song JY, Cheong HJ, Lee J, Woo HJ, Wie SH, Lee JS, Kim SW, Noh JY, Choi WS, Kim H, Kim KH, Kim WJ. Immunogenicity and safety of a cell culture-derived inactivated trivalent influenza vaccine (NBP607): A randomized, double-blind, multi-center, phase 3 clinical trial. Vaccine. 2015 Oct 5;33(41):5437-5444. doi: 10.1016/j.vaccine.2015.08.030. Epub 2015 Aug 24. PMID 26314625